CLINICAL TRIAL: NCT05558683
Title: Effect of the Vojta Therapy on Lipid Biomarkers Related to Myelin in Subjects With Multiple Sclerosis.
Brief Title: Effect of the Vojta Therapy in Patients Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aymara Abreu Corrales (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Sponsor-Investigator, Aymara Abreu Corrales, Principal investigator, Instituto de Neurociencia de Castillas y Leon
Organization: Instituto de Neurociencia de Castillas y Leon (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: MultipleSclerosisVojta
Record Dates: First submitted 2022-04-15; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
Keywords: Vojta Therapy; Bobath Therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Randomized Controlled Trials as Topic

STUDY DESIGN:
Intervention Model Description: Our study will be a Randomized Clinical Trial. It will be held at the Aymara Abreu Physiotherapy Clinic center, with a maximum duration of 1 year. It will consist of two parts. In the first stage of the treatment we will carry out an initial assessment, and in the second stage a final assessment. After that, the corresponding data analysis will be carried out.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Our population will be subjects diagnosed with MS. Prior to the study, the informed consent will be presented to the subjects. Said confidentiality will be contemplated in Organic Law 15/99 of December 13 on the Protection of personal data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vojta Reflex Locomotion Therapy (Active Comparator): The Vojta Method or Vojta Reflex Locomotion Therapy (TLRV) is a rehabilitative method for neuromusculoskeletal pathologies widely used in Europe. Its development is based on the concept of motor ontogenesis and tries to trigger innate motor reactions (reflex locomotion patterns) in the trunk and limbs from defined tactile and proprioceptive stimuli, starting from certain postures. This therapy presents differential elements with respect to other existing therapies, both for neurophysiological principles and for methodological principles. It is an active therapy, in which great concentration is required on the part of the patient, that is, both therapist and patient are the central axes of the treatment.
  Interventions: Other: Randomized clinical trial.
- Bobath Method (Active Comparator): Within physiotherapy, the Bobath concept is a valid and recognized option in the treatment of patients with neurological disorders, and therefore, of those diagnosed with MS. It was developed by Karel and Berta Bobath. The Bobath concept is defined as a problem-solving approach in the assessment and treatment of people with impaired neuromotor function, becoming a valid tool as part of the comprehensive treatment of people with MS
  Interventions: Other: Randomized clinical trial.

INTERVENTIONS:
Other: Randomized clinical trial. — Our study will be a Randomized Clinical Trial. It will be held at the Aymara Abreu Physiotherapy Clinic center, with a maximum duration of 1 year. It will consist of two parts. In the first stage of the treatment we will carry out an initial assessment, and in the second stage a final assessment. After that, the corresponding data analysis will be carried out.

SUMMARY:
Multiple sclerosis is the most common disabling neurological disease in young adults. Inflammation, demyelination, neurodegeneration, gliosis and repair processes are involved in its process, which are responsible for the heterogeneity and individual variability in the expression of the disease, the prognosis and the response to treatment. Clinically, MS manifests itself with the following symptoms: sensory focus, motor focus, spasticity, balance disorders, visual disturbances such as loss of vision or double vision or sphincter dysfunction.

The main subtypes of MS are relapsing-remitting, secondary progressive, primary progressive, and progressive relapsing. Clinically, RRMS presents the initial inflammatory phase, characterized by reversible flares with neurological dysfunction, followed by periods of remission. Approximately 40-50% of these patients progress to SPMS, where the disease gradually progresses from intermittent flare-ups to steadily progressive worsening, resulting in permanent disability due to massive axonal loss. PPMS is the most severe subtype, affecting approximately 10% of all cases, and manifesting as progressive degeneration without any remission.

DETAILED DESCRIPTION:
From the field of Physiotherapy, one of the main tools for the treatment of MS is physical exercise. Numerous studies show that exercising is safe and beneficial in people with MS, as long as it is done correctly and supervised by health professionals. Physical exercise is considered an important part of symptomatic and supportive treatment for people with MS, since it induces improvement of physiological functions affected by lack of physical activity and helps to manage some symptoms, such as spasticity, fatigue and lack of balance There are therapies within Physiotherapy that help treat MS such as the Vojta Method and the Bobath Method.

ELIGIBILITY:
Inclusion criteria:

* Persons with MS who have signed the informed consent.
* Persons of both sexes.
* Ages between 20 and 65 years.
* Subjects of both sexes diagnosed with multiple sclerosis on the EDSS (Expanded Disability Status Scale).

Exclusion criteria:

* Persons with multiple sclerosis with EDSS scale score equal to or greater than 7.0.
* Occurrence of a flare during the period of the patient's participation in the study.
* Pregnant women.
* Oncology patients.
* Non-acceptance and non-signing of informed consent.
* Refusal to participate in the study.
* Patients with severe cognitive impairment that does not allow them to understand the development of the study.
* Patients with cardiovascular instability.
* Patients who do not complete at least 75% of the scheduled sessions. Patients who do not present any of the contraindications contemplated for Vojta therapy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Respiratory function | 5 minutes
  Respiratory function will be assessed with a pressure manometer to measure peak inspiratory pressure.
Spasticity | 10 minutes
  Spasticity will be measured using the Tardieu scale.
Balance | 10 minutes
  The balance will be measured through the Berg scale.
Age | 1 minutes
Time reaction | 5 minutes
  Reaction time will be measured by the Cognifit test

SECONDARY OUTCOMES:
Myelin | 15 minutes
  Myelin will be me measured trough the tear duct whit phospholipid test strips

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abreu-Corrales A, Velasco A, Cuesta-Gomez A, Sanchez-Gonzalez JL. Impact of reflex locomotion and the Bobath concept on clinical and biomolecular parameters in people with multiple sclerosis: study protocol for a randomized controlled trial. Front Neurol. 2023 Aug 4;14:1209477. doi: 10.3389/fneur.2023.1209477. eCollection 2023. PMID 37602251